CLINICAL TRIAL: NCT01081613
Title: Imaging the Effect of HSP90 Inhibitor AUY922 on VEGF by Means of 89Zr-bevacizumab PET
Brief Title: Imaging HSP90 Inhibitor AUY922 on VEGF-89ZR-bevacizumab Positron Emission Tomography (PET)
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, PhD, University Medical Center Groningen
Other Study IDs: CAUY922A2101; 2008-005752-25 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: heat shock protein; breast cancer; PET imaging; bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — 89Zr-bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AUY922: Patients with estrogen receptor (ER) positive, hormone therapy refractory breast cancer.
  Interventions: Other: 89Zr-bevacizumab PET imaging

INTERVENTIONS:
Other: 89Zr-bevacizumab PET imaging — injection 89Zr-bevacizumab and 89 Zr-bevacizumab PET scan
  Other Names: 89Zr-bevacizumab

SUMMARY:
Inhibition of Heat Shock Protein (HSP)90 is a new, promising treatment modality for cancer patients, particularly in the setting of resistance. A reliable read out system (biomarker) for the evaluation of early treatment effect is of great importance in the development of this treatment modality, and could contribute to customize this treatment for individual patients. So far, no reliable biomarker has been described for HSP90 effect. Visualizing the effect of HSP90 on vascular endothelial growth factor (VEGF) secretion in vivo in the patient, by whole body 89Zr-bevacizumab uptake, can be of great importance in this respect, and may contribute to tailored made cancer treatment. The purpose of the present study is to evaluate the effect of HSP90 inhibition by AUY922 on VEGF by means of 89ZR-bevacizumab PET.

DETAILED DESCRIPTION:
This feasibility study is designed as a side study to the multicenter, international phase I-II trial with HSP90 inhibitor AUY922 (protocol CAUY922A2101), as part of the biomarker assessment. In protocol CAUY922A2101, section 4, the design of this phase I-II trial is described (p37, 38). Briefly, a dose-escalation study is performed according to phase I design in adult patients with advanced solid malignancies. This part is followed by a dose-expansion study according to a phase II design. In the latter part, breast cancer patients are enrolled that are either refractory to hormone- or trastuzumab treatment (both treatment arms, n=40 patients), on the maximal tolerated dose of AUY922 based on the phase I part of the study. Patients with ER positive, hormone therapy refractory breast cancer, will receive a 89Zr-bevacizumab PET scan as part of the present side study protocol, which will be performed in collaboration with the Royal Marsden Hospital (United Kingdom).

To this end, a 89Zr-bevacizumab PET scan will be performed before (baseline) and during treatment with HSP90 inhibitor AUY922, as described below.

A minimum of six patients will be entered to evaluate whether the effect of HSP90 inhibition by AUY922 can be detected with a 89Zr-bevacizumab PET scan

ELIGIBILITY:
Inclusion Criteria:

* patients with ER positive, hormone therapy refractory breast cancer
* participation in the phase I-II trial with HSP90 inhibitor AUY922 (in- and exclusion criteria for the study with AUY922 are described in protocol CAUY922A2101, Clinical Trials no NCT00526045A.

Exclusion Criteria:

* no participation in the phase I-II trial with HSP90 inhibitor AUY922

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ER positive, hormone therapy refractory breast cancer, who are participating in the phase I-II trial with HSP90 inhibitor AUY922
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of HSP90 inhibition by AUY922 on VEGF by means of 89Zr-bevacizumab PET. | 2 years
  Primary endpoint: measurement of decreased VEGF compared to baseline. A decline is defined as a decrease of at least 30% in mean Standardized Uptake Value (SUV) in a maximum of three lesions.

CONTACTS AND LOCATIONS:
Overall Officials: C.P. Schröder, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands